CLINICAL TRIAL: NCT01454908
Title: Investigation of Unicompartmental Knee Arthroplasty and Functional, Daily Activities: A Quantitative Assessment of Gait, Sit-to-Stand, and Stair Climbing
Brief Title: Oxford Partial Knee Kinematics Gait Analysis Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The CORE Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100-U-005; NCT00576966 (obsolete NCT alias)
Record Dates: First submitted 2011-10-13; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Medial Knee Compartment Arthritis
Keywords: partial knee arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Partial Knee Arthroplasty (Other): Oxford Mobile Bearing Unicompartmental Knee Arthroplasties
  Interventions: Device: Oxford Partial Knee

INTERVENTIONS:
Device: Oxford Partial Knee — The Oxford partial knee contains tibial and medial components and a mobile meniscal bearing.

SUMMARY:
The objective of this study is to compare the effect on gait of unicompartmental knee arthroplasty (UKA), using the Oxford Partial Knee, versus normal knee.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medial knee compartment arthritis

Exclusion Criteria:

* Patients with diagnoses other than osteoarthritis (i.e., rheumatoid arthritis, psoriatic arthritis, etc.)
* Patients with significant diseases of other joints of the lower extremity
* Patients with a diagnosed disorder with gait disturbance (e.g. lower extremity weakness, prior lower extremity arthrodesis, diagnosed movement disorders, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-04; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score (KSS) | up to 1 month pre-operatively and at 1 year post operatively

SECONDARY OUTCOMES:
Range of Motion (ROM) | up to 1 month pre-operatively and at 1 year post operatively

CONTACTS AND LOCATIONS:
Locations (1):
- SHRI-CORE Orthopedic Research Lab, Sun City West, Arizona, United States